CLINICAL TRIAL: NCT05293041
Title: Influence of Argipressin on Blood Loss During Hepatic Resection; a Double-blinded, Randomized Placebo-controlled Trial (ARG-01)
Brief Title: Argipressin's Influence on Blood Loss During Hepatic Resection
Acronym: ARG-01
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kristina Svennerholm (Other)
Responsible Party: Sponsor-Investigator, Kristina Svennerholm, Principal investigator, MD, PhD, Sahlgrenska University Hospital
Organization: Sahlgrenska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARG-01
Record Dates: First submitted 2021-11-15; First posted 2022-03-24 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Colon Cancer Liver Metastasis; Inflammatory Response; Vasopressin Causing Adverse Effects in Therapeutic Use
Keywords: hepatic surgery; vasopressin; liver surgery; colon cancer metastasis; transfusion; blood loss; inflammatory response; pain; coagulation
MeSH Terms: conditions — Diabetes Insipidus; Hemorrhage; Pain; Thrombosis | interventions — Arginine Vasopressin; Arginine

STUDY DESIGN:
Intervention Model Description: Singel center double-blinded, randomized, placebo-controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomisation will be handled by a nurse not involved in the study, and both the patient, treating physician and nurse, the study nurse and the investigators will be blinded to the study treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Argipressin (Experimental): Patients will be treated with Empressin® 0.8 U/ml, 0.056 ml/kg/h during surgery.
  Interventions: Drug: Argipressin
- Placebo (Placebo Comparator): Patients will receive normal saline 0.056 ml/kg/h during surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Argipressin — Infusion of Argipressin 0.8 U/ml, 0.056 ml/kg/h will be started as soon as the central line is placed, and continued until the end of surgery in the treatment arm.
  Other Names: Arg
  Arms: Argipressin
Drug: Placebo — Infusion of Normal Saline 0.056 ml/kg/h will be started as soon as the central line is placed, and continued until the end of surgery in the placebo arm.
  Other Names: control
  Arms: Placebo

SUMMARY:
Infusion of Argipressin during hepatic resection surgery may reduce blood loss. It may also reduce transfusion requirements, and mitigate the perioperative inflammatory response compared to placebo. Subjects will be randomized to infusion of Argipressin or placebo during surgery. Blood loss, transfusion requirements, surgical data including length of stay in hsopital, inflammatory markers and markers of renal- intestinal- and cardiac injury will be assessed. Two sub-studies has been added; one for evaluation of coagulation function, and one for assessment of pain scores and morphine consumption.

DETAILED DESCRIPTION:
Hepatic resection is a major surgical intervention with high risk of substantial blood loss. The surgical means to reduce blood loss may impair perfusion and induce intestinal congestion. If blood flow to the liver can be influenced by pharmacological means, blood loss and transfusion requirements may be reduced. Moreover, the inflammatory system is involved in cancer development, and the anti-inflammatory properties of Argipressin may decrease the inflammatory response after hepatic surgery.

Argipressin is an endogenous substance, and part of the body's response to stress and trauma. Argipressin affects V1-receptors to produce vasoconstriction. It is also involved in inflammatory reactions and affects platelets.

Patients will be stratified according to planned type of surgery (open/laparoscopic) and planned extent of resection, and randomized to etiher infusion of Argipressin or placebo (normal saline) during surgery. In all other aspects, the participants will be treated according to the institution protocol for hepatic resection. The study drug will be started as soon as the central line is placed, and discontinued at the end of surgery. Hemodynamic data will be collected during surgery, and blood and urine-samples will be obtained during and after surgery for analysis of inflammatory markers and markers of organ injury.

ELIGIBILITY:
Inclusion Criteria:

1. Participant planned for hepatic resection (open or laparoscopic, regardless of indication for surgery).
2. Age ≥18 years.
3. ASA class I-III.
4. Signed informed consent form

Exclusion Criteria:

1. Participant does not understand the given information, and/ or cannot give written informed consent.
2. Simultaneous operation of tumor with other localization, or surgery for superficial single hepatic tumor less than 2 cm, expected to be of short duration and with minimal blood loss.
3. Terminal kidney failure (estimated preoperative GFR< 15 ml/min)
4. Pregnancy or lactation.
5. Known allergy to Empressin®.
6. Patient included in other interventional study, interacting with the endpoints in the present study, or previous randomization in this study.
7. Hyponatremia (S-Na < 130 mmol/L)
8. Patient considered ineligible for other surgical or medical reason.
9. Present infection. Patients with systemic inflammatory disease, inflammatory bowel disease or preoperative corticosteroid treatment will not be eligible for the subgroups where cytokines and interleukins are investigated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2022-03-27 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Blood loss | through surgery, an average of 8 hours
  Blood loss at the end of surgery, measured according to the investigator's instructions, by visual assessment of suction devises and gauze, and subtraction of ascites and irrigation fluids.

SECONDARY OUTCOMES:
Blood transfusion | At end of surgery and until postoperative day 2 or 5 respectively
  Blood transfusion (ml) at the end of surgery and at postoperative day 1 and 2 and 5 respectively.
Inflammatory markers-regular | Measured throughout the study until postoperative day 2 (laparoscopic resection) or postoperative day 5 (open resection)
  Levels of White Blood Cell count, C Reactive Protein, Platelet count and Albumin at the end of surgery and postoperative day 1-5
Inflammatory markers- extended | Measured at throughout the study until postoperative day 2.
  Levels of Interleukin (IL)-1 Beta, IL-6, IL-8, IL-10, Monocyte chemoattractant protein-1, Stromal Cell-Derived Factor-1 alpha, Intercellular Adhesion Molecule, Complement (C) 3a, C5b-9 at the end of surgery and postoperative day 1 and 2.
surgical data | at the end of surgery, approximately 5 hours after start of surgery
  duration of Pringles manouvre (min), duration of resection phase (min) and surgery (min)
Tranexamic Acid | at the end of surgery, approximately 5 hours after start of surgery
  use of tranexamic acid (mg)
CVP (anesthesiological data) | during surgery
  achievement of CVP (central venous pressure) goal (mmHg), as recorded on the Phillips monitor.
Noradrenaline use (anesthesiologigal data) | during surgery
  Total use of noradrenaline (micrograms/minutes of surgery/ bodyweight)
use of diuretics | until postoperative day 1
  Furosemide use (mg)
urine output | until postoperative day 1
  urine output (ml)
postoperative complications | 30 days after surgery
  Postoperative complications including death and radicality of resection at 30-day follow up.
Length of stay | From admission in hospital to discharge, expected time 2-5 days but will be followed until actual discharge, which may be several months.
  Length of stay in hospital
Plasma Creatinine (change in organ damage markers) | from baseline (before surgery) to postoperative day 2 and 5 respectively.
  Change in plasma creatinine (micro-mole/L)
Urine samples (change in organ damage markers) | from baseline to end of surgery, approximately 5 hours
  Change in urine creatinine and urine [TIMP-2] x [IGFBP-7] (quota, no unit)
Cardiac marker (change in organ damage markers) | from baseline to postoperative day 1
  Change in hs- TNI (ng/L)
Lactate (change in organ damage markers) | from baseline to postoperative day 1
  change in plasma lactate
I-FABP (change in organ damage markers) | from baseline to postoperative day 1
  Change in I-FABP (ng/L)

OTHER OUTCOMES:
oral morphine eqivalents | from day of surgery, postoperative day 1,2 and at discharge from hospital (but no longer than post operative day 5)
  total opioid consumption converted to oral morphine eqivalents (mg)
Numeric Rating Scale (NRS) | Once daily at day of surgery, postoperative day 1 and 2
  pain assement by Numeric Rating Scale 0-10 (0= no pain, 10= worst pain imaginable), at rest and at activity
Clotting Time (CT) | before anesthesia, at end of surgery (assessed up to one hour after closing of the abdomen) and postoperative day 1
  Clotting Time (CT) measured by ROTEM (Thrombelastometry) in Extem, Intem, Fibtem, Heptem channels
Clot Formation time (CFT) | before anesthesia, at end of surgery (assessed up to one hour after closing of the abdomen) and postoperative day 1
  Clot Formation time (CFT) measured by ROTEM (Thrombelastometry) in Extem, Intem, Fibtem, Heptem channels
Amplitude at 10 minutes (A10) | before anesthesia, at end of surgery (assessed up to one hour after closing of the abdomen) and postoperative day 1
  Amplitude at 10 minutes (A10) measured by ROTEM (Thrombelastometry) in Extem, Intem, Fibtem, Heptem channels
Maximum Clot Firmness (MCF) | before anesthesia, at end of surgery (assessed up to one hour after closing of the abdomen) and postoperative day 1
  Maximum Clot Firmness (MCF) measured by ROTEM (Thrombelastometry) in Extem, Intem, Fibtem, Heptem channels
vWf | before anesthesia, at end of surgery (assessed up to one hour after closing of the abdomen) and postoperative day 1
  von Willebrand factor (vWf)
fVIII | before anesthesia, at end of surgery (assessed up to one hour after closing of the abdomen) and postoperative day 1
  factor VIII

CONTACTS AND LOCATIONS:
Overall Officials: kristina svennerholm, MD PhD, Principal Investigator — Senior Consultant Anesthesia and Intensive Care, Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Metadata will be shared by the Swedish National Data Service (SND, https://snd.gu.se/en) and selected psedonymised data will be made available on reasonable request, after proper confidentiality and ethics assessment. The extent of data made available will be decided after study closure, and also the time span for availability.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months after study closure, and maximum 25 years
Access Criteria: Confidentiality and ethics assessment.
URL: https://snd.gu.se/en

REFERENCES:
- [Derived] Wisen E, Pivodic A, Skagervik A, Rizell M, Bown LS, Ricksten SE, Svennerholm K. Argipressin for prevention of blood loss in hepatic resection: a randomised, placebo-controlled, double-blind trial. Br J Anaesth. 2025 Oct 30:S0007-0912(25)00672-5. doi: 10.1016/j.bja.2025.09.021. Online ahead of print. PMID 41173775
- [Derived] Wisen E, Kvarnstrom A, Sand-Bown L, Rizell M, Pivodic A, Ricksten SE, Svennerholm K. Argipressin for prevention of blood loss during liver resection: a study protocol for a randomised, placebo-controlled, double-blinded trial (ARG-01). BMJ Open. 2023 Aug 24;13(8):e073270. doi: 10.1136/bmjopen-2023-073270. PMID 37620260

DOCUMENTS (2):
  • Study Protocol (2025-02-28): https://cdn.clinicaltrials.gov/large-docs/41/NCT05293041/Prot_002.pdf
  • Statistical Analysis Plan (2023-02-27): https://cdn.clinicaltrials.gov/large-docs/41/NCT05293041/SAP_001.pdf